CLINICAL TRIAL: NCT03386279
Title: A PHASE 1, RANDOMIZED, PLACEBO-AND POSITIVE-CONTROLLED CROSSOVER STUDY TO DETERMINE THE EFFECT OF SINGLE-DOSE PF-04965842 ON QTC INTERVAL IN HEALTHY VOLUNTEERS
Brief Title: A Study To Determine The Effect Of Single-dose PF-04965842 On QTc Interval In Healthy Volunteers Compared With Placebo and Moxifloxacin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: B7451027; 2017-004472-61 (EudraCT Number)
Record Dates: First submitted 2017-12-21; First posted 2017-12-29 (Actual); Last update posted 2019-10-14 (Actual); Status verified 2019-10

CONDITIONS: Healthy Volunteers
Keywords: healthy volunteers
MeSH Terms: interventions — abrocitinib; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: PF-04965842 and placebo oral tablets will be prepared in the CRU by 2 operators, 1 of whom is an unblinded pharmacist. PF-04965842 and placebo will be administered in blinded fashion to the subject.
  Moxifloxacin 400 mg tablets will be packaged in an open-label manner at the CRU in the individual dosing containers by 2 operators, 1 of whom is an appropriately qualified and experienced member of the study staff (eg, physician, nurse, physician's assistant, practitioner, or pharmacist).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Sequence 1 (Other): Sequential allocation to PF-04965842 600 mg (oral, single dose), placebo (oral, single dose), and moxifloxacin 400 mg (oral, single dose)
  Interventions: Drug: PF-04965842; Drug: Moxifloxacin; Drug: Placebo
- Sequence 2 (Other): Sequential allocation to PF-04965842 600 mg (oral, single dose), moxifloxacin 400 mg (oral, single dose), and placebo (oral, single dose)
  Interventions: Drug: PF-04965842; Drug: Moxifloxacin; Drug: Placebo
- Sequence 3 (Other): Sequential allocation to placebo (oral, single dose), PF-04965842 600 mg (oral, single dose), and moxifloxacin 400 mg (oral, single dose).
  Interventions: Drug: PF-04965842; Drug: Moxifloxacin; Drug: Placebo
- Sequence 4 (Other): Sequential allocation to placebo (oral, single dose), moxifloxacin 400 mg (oral, single dose), and PF-04965842 600 mg (oral, single dose)
  Interventions: Drug: PF-04965842; Drug: Moxifloxacin; Drug: Placebo
- Sequence 5 (Other): Sequential allocation to moxifloxacin 400 mg (oral, single dose), PF-04965842 600 mg (oral, single dose), and placebo (oral, single dose)
  Interventions: Drug: PF-04965842; Drug: Moxifloxacin; Drug: Placebo
- Sequence 6 (Other): Sequential allocation to moxifloxacin 400 mg (oral, single dose), placebo (oral, single dose) and PF-04965842 600 mg (oral, single dose)
  Interventions: Drug: PF-04965842; Drug: Moxifloxacin; Drug: Placebo

INTERVENTIONS:
Drug: PF-04965842 — one single dose of 600 mg by mouth
Drug: Moxifloxacin — one single dose of 400 mg by mouth
Drug: Placebo — one single dose by mouth

SUMMARY:
This is a Phase 1, single-dose, randomized, 3-treatment, 3-period cross-over, sponsor-open, placebo-and positive-controlled trial to be conducted in approximately 36 adult healthy volunteers. There will be 3 crossover treatments: PF-04965842 600 mg (A), placebo (B) and moxifloxacin 400 mg (C). Treatment assignments to PF-04965842 and placebo will be blinded to the subjects, investigator and Clinical Research Unit (CRU) staff (except pharmacist) but open to the sponsor. Moxifloxacin administration will be unblinded. Dosing in each of the 3 treatment periods will be separated by a washout period of at least 5 days

Screening evaluation will occur within the 28 days prior to dosing in the first treatment period. During each treatment period, eligible subjects who meet the entry criteria will be admitted on Day -1, prior to treatment administration on Day 1, and will reside in the CRU until completion of protocol assessments on Day 2. There will be a washout of at least 5 days between dose administrations in consecutive crossover treatment periods. After completion of the 3 study periods or upon withdrawal from the study, subjects will return for a follow-up visit approximately 7-14 days following last dose of investigational product. Further follow-up contact will be made at least 28 calendar days and up to 35 calendar days after the last administration of the investigational product to capture any potential AEs and concomitant treatments, and to confirm appropriate contraception usage, contact with the subject may be done via phone. For each subject, the duration of participation from Day 1 admission to follow-up visit will be approximately 10 weeks. The follow-up call will occur up to 4 weeks after the follow-up visit.

In each treatment period, the subject will be admitted to the CRU the day prior to dosing. Genotyping samples for CYP2C19 and CYP2C9 will be collected pre-dose in Period 1 only. The subject will receive a single dose of the assigned trial medication in the morning of Day 1. Triplicate 12-lead ECG measurements (approximately 2 minutes apart) will be performed on Days 1 and 2 of each treatment period as follows: -1, -0.5 and 0 hours pre-dose and at 0.25, 0.5, 1, 2, 3, 6, 12, and 24 hours post-dose. Blood samples will be collected following the 0 hour and post-dose ECG measurements at the same time-points to evaluate the PK of PF-04965842 and moxifloxacin (if needed). Clinical safety laboratory tests will be performed on Day -1 and at 24 hours on Day 2, and vital signs (supine pulse rate and BP) will be monitored pre-dose and at 2 and 6 hours post-dose on Day 1 and at 24 hours on Day 2. The subject will be discharged from the CRU after completing all trial procedures of the particular treatment period in the morning of Day 2 (24 hours post-dose).

ELIGIBILITY:
Inclusion Criteria:

1. Healthy female subjects of nonchildbearing potential and/or male subjects who, at the time of screening, are between the ages of 18 and 55 years, inclusive. Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including BP and pulse rate measurement, 12-lead

   ECG, or clinical laboratory tests. Female subjects of nonchildbearing potential must meet at least 1 of the following criteria:
   1. Achieved postmenopausal status, defined as follows: cessation of regular menses for at least 12 consecutive months with no alternative pathological or physiological cause; status may be confirmed with a serum follicle-stimulating hormone (FSH) level confirming the postmenopausal state;
   2. Have undergone a documented hysterectomy and/or bilateral oophorectomy;
   3. Have medically confirmed ovarian failure. All other female subjects (including female subjects with tubal ligations) are considered to be of childbearing potential.
2. Body mass index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lb).
3. Evidence of a personally signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the study.
4. Subjects who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria:

1. Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic (including alcoholic liver disease, nonalcoholic steatohepatitis (NASH), autoimmune hepatitis, and hereditary liver diseases), psychiatric, neurological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
2. Evidence or history of clinically significant dermatological condition (eg, contact dermatitis or psoriasis) or visible rash present during physical examination.
3. Subjects, who according to the product label for moxifloxacin, would be at increased risk if dosed with moxifloxacin (ie, including but not limited to subjects with history of myasthenia gravis, tendinitis/tendon rupture).
4. Self-reported history or risk factors for QT prolongation or torsades de pointes (eg, organic heart disease, congestive heart failure, hypokalemia, hypomagnesaemia, congenital long QT syndrome, myocardial ischemia or infarction), congenital deafness, family history of sudden death, and family history of long QT syndrome.
5. Any condition possibly affecting drug absorption (eg, gastrectomy).
6. A positive urine drug test.
7. History of regular alcohol consumption exceeding 14 drinks/week for female subjects or 21 drinks/week for male subjects (1 drink = 5 ounces [150 mL] of wine or 12 ounces [360 mL] of beer or 1.5 ounces [45 mL] of hard liquor) within 6 months before screening.
8. Treatment with an investigational drug within 30 days (or as determined by the local requirement) or 5 half-lives preceding the first dose of investigational product (whichever is longer).
9. Subjects with known prior participation (ie, randomized and received at least 1 dose of investigational product) in a trial involving PF-04965842.
10. Screening supine systolic BP <90 mm Hg or <140 mm Hg following at least 5 minutes of supine rest OR Screening supine diastolic BP <50 mm Hg or <90 mm Hg following at least 5 minutes of supine rest. If a subject meets any of these criteria, the BP should be repeated 2 more times and the average of the 3 BP values should be used to determine the subject's eligibility.
11. Screening supine 12-lead ECG demonstrating: QTcF >450 msec OR QRS interval >120 msec. If QTcF exceeds 450 msec, or QRS exceeds 120 msec, the ECG should be repeated 2 more times and the average of the 3 QTcF or QRS values should be used to determine the subject's eligibility.
12. Subjects with ANY of the following abnormalities in clinical laboratory tests at screening, as assessed by the study-specific laboratory and confirmed by a single repeat test, if deemed necessary:

    Aspartate aminotransferase (AST)/serum glutamic oxaloacetic transminase (SGOT) or alanine aminotransferase (ALT)/serum glutamic pyruvic transminase (SGPT) <1.5 × upper limit of normal (ULN).

    Total bilirubin level 1.5 × ULN; subjects with a history of Gilbert's syndrome may have direct bilirubin measured and would be eligible for this study provided the direct bilirubin level is ULN.
13. Known relevant history of elevated liver function tests (LFTs).
14. History of tuberculosis (TB) or active or latent or inadequately treated infection.
15. Fertile male subjects who are unwilling or unable to use a highly effective method of contraception as outlined in this protocol for the duration of the study and for at least 28 days after the last dose of investigational product.
16. Use of prescription or nonprescription drugs and dietary supplements within 7 days or 5 half-lives (whichever is longer) prior to the first dose of investigational product. As an exception, acetaminophen/paracetamol may be used at doses of 1g/day. Limited use of nonprescription medications that are not believed to affect subject safety or the overall results of the study may be permitted on a case-by-case basis following approval by the sponsor. Herbal supplements and hormone replacement therapy must have been discontinued at least 28 days prior to the first dose of investigational product.
17. Use of tobacco- or nicotine- containing products in excess of the equivalent of 5 cigarettes per day.
18. Blood donation (excluding plasma donations) of approximately 1 pint (500 mL) or more within 60 days prior to dosing.
19. History of hypersensitivity, allergy, severe adverse drug reaction or intolerance to quinolone antibiotics, including moxifloxacin.
20. History of human immunodeficiency virus (HIV), hepatitis B, or hepatitis C; positive testing for HIV, hepatitis B surface antigen (HepBsAg), hepatitis B core antibody (HepBcAb), or hepatitis C antibody (HCVAb). As an exception, a positive hepatitis B surface antibody (HepBsAb) finding as a result of subject vaccination is permissible.
21. Unwilling or unable to comply with the criteria in the Lifestyle Requirements section of this protocol.
22. Subjects who are investigator site staff members directly involved in the conduct of the study and their family members, site staff members otherwise supervised by the investigator, or subjects who are Pfizer employees, including their family members, directly involved in the conduct of the study.
23. Other acute or chronic medical or psychiatric condition including recent (within the past year) or active suicidal ideation or behavior or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2018-07-02 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2018-10-01 (Actual)

PRIMARY OUTCOMES:
Relationship between QTc change (msec) and PF-04965842 concentration | Zero hour (prior to zero hour treatment administration), and at 0.25, 0.5, 1, 2, 3, 6, 12 and 24 hours post-dose
  Linear mixed effects modeling will be derived from ECGs and PK blood samples at the stated time points with an aim to demonstrate the lack of effect on QTc interval in healthy volunteers, of a supra-therapeutic concentration after administering a dose of 600 mg PF-04965842 compared with placebo.

SECONDARY OUTCOMES:
Relationship between QTc change (msec) and PF-04965842 concentration | Zero hour (prior to zero hour treatment administration), and at 0.25, 0.5, 1, 2, 3, 6, 12 and 24 hours post-dose
  Linear mixed effects modeling will be derived from ECGs and PK blood samples at the stated time points. with an aim to demonstrate the lack of effect on QTc interval in healthy volunteers, of a therapeutic concentration after administering a dose of 600 mg PF-04965842 compared with placebo.
Time matched mean differences in QTc between moxifloxacin and placebo | Zero hour (prior to zero hour treatment administration), and 0.25, 0.5, 1, 2, 3, 6, 12 and 24 hours post-dose
  Time matched mean differences in QTc between moxifloxacin and placebo at each post dose time point, including at the historical moxifloxacin Tmax of 3 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Clinical Research Unit, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Wojciechowski J, Malhotra BK, Wang X, Fostvedt L, Valdez H, Nicholas T. Population Pharmacokinetics of Abrocitinib in Healthy Individuals and Patients with Psoriasis or Atopic Dermatitis. Clin Pharmacokinet. 2022 May;61(5):709-723. doi: 10.1007/s40262-021-01104-z. Epub 2022 Jan 21. PMID 35061234
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B7451027